CLINICAL TRIAL: NCT03614572
Title: Advancing Adolescent Bedtime by Using Motivational Interviewing and Text Reminders - A Randomized Controlled Trial
Brief Title: Advancing Adolescent Bedtime by MI and Text Reminders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN NGAN YIN, Research Associate, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15163071
Record Dates: First submitted 2018-07-21; First posted 2018-08-03 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Sleep Deprivation
Keywords: Sleep deprivation; Motivational Interviewing; Text reminders
MeSH Terms: conditions — Sleep Deprivation | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor will be blinded to the condition of the subjects
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group MI (Experimental): The structure and content of the active intervention programme will be developed and adopted on the basis of previous research on sleep educational programme and motivational interviewing techniques. The whole treatment package consists of 4 sessions of group therapy (n=6-8) followed by 3 week daily text reminders.
  Interventions: Behavioral: Group MI
- Control group (No Intervention): Control group will no receive any intervention

INTERVENTIONS:
Behavioral: Group MI — refer to the arm description
  Other Names: Motivational interviewing
  Arms: Group MI

SUMMARY:
Chronic sleep deprivation among adolescents is a prevalent health problem across the world and is associated with a series of short and long term consequences. However, effective interventions targeting on this vulnerable adolescent population is very limited. Majority of the previous sleep education programme are conducted in a school context which personal factors and individualized problems were not addressed. In addition, failure to address "knowledge-action gap" may also explain why individual fail to enact health behaviors even holding positive motivation. In regard to this, investigators proposed an active and person-oriented protocol with the aid of advanced technology in order to improve adolescent sleep health.

DETAILED DESCRIPTION:
This study will conduct a randomized control trial to evaluate the effectiveness of group-based sleep intervention using motivational interviewing plus text reminders in changing adolescent sleep deprivation problem with both subjective and objective measurements. The intervention will consists of 4 weekly group therapy targeting on adolescent with school day sleep duration less than 7 hours.

ELIGIBILITY:
Inclusion Criteria:

* Chinese aged 12-18 years old
* Written informed consent of participation into the study is given by adolescents and his/her parents;
* Being able to comply with the study protocol;
* Having weekday sleep duration less than 7 hours for past 1 month as reported by questionnaire and average of <7hr weekday sleep as reported by sleep diary as an indication of chronic sleep deprivation status.
* Possess a mobile phone

Exclusion Criteria:

* A current or past history of neuropsychiatric disorder(s);
* A prominent medical condition or taking medication with potential side effects that may influence sleep quantity and quality
* Having a clinical sleep disorder that may potentially contribute to the disruption of sleep quantity and quality as ascertained by both Structured Diagnostic Interview for Sleep patterns and Disorders such as insomnia, delayed sleep phase and narcolepsy.
* have enrolled in any intervention programme that may affect their sleep patterns in the past three months or are planning to join intervention programme in the next three month

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 212 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Change of Sleep duration by sleep diary | Baseline, 1 week, 3 month and 6 month after treatment
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: total sleep time (TST) in hours
Change of Sleep duration by actigraphy | Baseline, 1 week, 3 month and 6 month after treatment
  Sleep parameter estimated by actigraphy: total sleep time (TST) in hours

SECONDARY OUTCOMES:
Change of Sleep knowledge | Baseline, 1 week, 3 month and 6 month after treatment
  Sleep knowledge is measured by Sleep Knowledge Questionnaire. It consists of 25 items, ranging from -50 to 50 with higher score indicates better sleep knowledge
Change of Daytime Sleepiness | Baseline, 1 week, 3 month and 6 month after treatment
  Paediatric Daytime Sleepiness Scale (PDSS) is an 8-item self-rated scale measuring daytime sleepiness, ranging in total scores from 0 to 32 with higher scores indicating more sleepiness.
Change of Quality of Life | Baseline, 1 week, 3 month and 6 month after treatment
  KIDSCREEN-27 health questionnaire for children and young people for the measurement of quality of life by rating 27 items related to general health on a 5 point Likert scale.
  There are five subscales on: physical well-being (possibly scored from 5 to 25), psychological well-being (possibly scored 7 to 35), autonomy & parents (possibly scored 7 to 35), peers & social support (possibly scored 4 to 20), and school environment (possibly scored 4 to 20). A grand total score can be calculated by summing up the five sub scores. In all cases, a higher score represents higher perceived well-being.
Change of Sleep Hygiene | Baseline, 1 week, 3 month and 6 month after treatment
  Adolescent Sleep Hygiene Scale (ASHS): It is a 28-item instrument used to assess how adolescent apply sleep hygiene practice. total score range from 28 to 168 with higher score indicates better sleep practice. The instrument assessed adolescent sleep practice in nine domains: physiological(5 items, score 5-30), cognitive(6 items, score: 6 to 36), emotional(3 items; score: 3-18), sleep environment(4 items; score: 4-24), daytime sleep(1 items; score 1-6), substance(2 items; score: 2 to 12), bedtime routine(1 items; score:1-6), sleep stability(4 items; score: 4 to 16) and bedroom sharing(2 items; score 2-12).
Change of Anxiety and depressive symptoms | Baseline, 1 week, 3 month and 6 month after treatment
  Hospital Anxiety and Depression Scale (HADS) is a self-assessed scale for detecting states of depression and anxiety. The depression subscale range in scores from 0 to 21, with higher scores indicating severer states of depression. Similarly, the anxiety subscale range in scores from 0-21 with higher scores indicating severer states of anxiety. No additional computation will be made with the two subscores.
Change of Academic performance | Baseline, 3 month and 6 month after treatment
  Academic performance is evaluated by the difference in average grade point between baseline, 3 month and 6 month.
Change of objective cognitive performance (inhibitory ability) | Baseline, 3 month and 6 month after treatment
  Go/No-go Task for assessing inhibitory ability. In Go/No-go Task, a higher error rate indicates lower inhibition control.
Change of objective cognitive performance (working memory by digit span) | Baseline, 3 month and 6 month after treatment
  Digit Span Task for assessing working memory capacity. In Digit Span Task, a higher number of recalled digits indicates better working memory.
Change of objective cognitive performance (working memory by N-Back) | Baseline, 3 month and 6 month after treatment
  N-back Task for assessing working memory capacity and manipulation. In N-back Task, a d prime score will be calculated based on the signal detection theory, where a higher score indicates better working memory performance.
Change of risk-taking & decision making | Baseline, 3 month and 6 month after treatment
  Balloon Analogue Risk Task for assessing risk-taking and decision-making. In Balloon Analogue Risk Task, a score will be calculated by averaging the number of pumps on unexploded blue balloons, where a higher score indicates more risk-taking and impulsive propensities.

CONTACTS AND LOCATIONS:
Overall Officials: Ngan Yin Chan, Mphi, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Psychiatry, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan NY, Chen SJ, Ngan CL, Li SX, Zhang J, Lam SP, Chan JWY, Yu MWM, Chan KCC, Li AM, Wing YK. Advancing adolescent bedtime by motivational interviewing and text message: a randomized controlled trial. J Child Psychol Psychiatry. 2025 Jul;66(7):1005-1017. doi: 10.1111/jcpp.14115. Epub 2025 Jan 20. PMID 39834005